CLINICAL TRIAL: NCT00360633
Title: Psychiatric and Cognitive Manifestations of Parkinson's Disease: A Prospective Cohort Study
Brief Title: Psychiatric and Cognitive Manifestations of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12-03082
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Impulse control disorder; Dopamine agonist withdrawal syndrome; Anxiety; Depression; Healthcare Utilization; Disability; Quality of life; Cognitive function; Psychosis; Apathy; Dyskinesias; Wearing off
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders; Anxiety Disorders; Depression; Psychotic Disorders; Lethargy; Dyskinesias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson's Disease (PD) is often thought of as affecting movement only. In fact, most patients also experience psychiatric and cognitive symptoms, sometimes from the disease itself, and sometimes as a side-effect of PD medications. The goals of this study are to evaluate the causes, effects, and clinical correlates of psychiatric and cognitive symptoms in PD.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is defined by the presence of motor symptoms, but in recent years there has been increasing recognition of non-motor manifestations, including anxiety, depression, and cognitive symptoms. In addition, PD medications have been shown to cause impulse control disorders, cognitive changes, and non-motor withdrawal symptoms (dopamine agonist withdrawal syndrome) when they are discontinued. The goals of this study are to test the hypothesis that the presence of psychiatric and cognitive symptoms are associated with greater self-perceived disability (out of proportion to objective deficits), increased utilization of healthcare resources, and decreased quality of life. In addition, we will examine the clinical correlates of these psychiatric symptoms. To test these hypotheses, we will screen PD patients for anxiety, depression, impulse control disorders, and dopamine agonist withdrawal syndrome, and compare cases and controls with regard to demographic characteristics, motor features of PD, disability, healthcare utilization, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease (or healthy control subject)
* Age >=21 and <=99
* Capacity to provide informed consent
* Ability to complete the questionnaires

Exclusion Criteria:

* Clinical diagnosis of dementia
* Terminal illness (life expectancy < 12 months)
* Presence of a neurodegenerative disorder other than Parkinson's Disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with Parkinson's Disease who are seen for their routine medical care at the NYU Parkinson's and Movement Disorders Center.
  2. Matched healthy control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-06; Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Non-motor symptom progression | Chronic

SECONDARY OUTCOMES:
Motor symptom progression | Chronic

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Nirenberg, MD, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- See also: NYU Parkinson's Disease and Movement Disorders Center — http://parkinson.med.nyu.edu/